CLINICAL TRIAL: NCT00778141
Title: A Relative Bioavailability Study of Metformin HCl 750 mg XR Tablets Under Non-Fasting Conditions.
Brief Title: Bioequivalence Study of Metformin HCl 750 mg XR Tablets Under Non Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B045503
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalecne metformin HC1 750 mg extended-release tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): metformin HC1 750 mg extended-release tablets
  Interventions: Drug: metformin HC1 750 mg extended-release tablets
- 2 (Active Comparator): Glucophage® XR 750 mg tablets
  Interventions: Drug: metformin HC1 750 mg extended-release tablets

INTERVENTIONS:
Drug: metformin HC1 750 mg extended-release tablets

SUMMARY:
The objective of this study is to compare the relative bioavailability of metformin HC1 750 mg extended-release tablets (Ranbaxy) with that of Glucophage® XR 750 mg tablets (Bristol Myers Squibb) in healthy, adult, subjects under non-fasting conditions.

DETAILED DESCRIPTION:
1. Design: Single dose, randomized, two-period, two-treatment, two- sequence crossover study under non-fasting conditions comparing equal doses of the test and reference products.
2. Interval between dosing periods: At least one week
3. Period of confinement: From at least 10.5 hours before dosing until after the 36 hour blood collection each period. Subjects will return to the clinic for subsequent blood collations.

A total of thirty six (36) subjects were enrolled in this study; 33 completed the study.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects selected for this study will be at least 18 years of age.
2. Each subject shall be given a general physical examination within 28 days of initiation of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history.
3. Each female subject will be given a serum pregnancy test as part of the pre-study screening process. At the end of the study, the subjects will have an exit evaluation consisting of interim history, global evaluation, and clinical laboratory measurements.
4. Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trial for clinical laboratory measurements.
5. Clinical laboratory measurements will include the hematology, clinical chemistry, urine analysis, HIV screening, Hepatitis B & C, drugs of abuse scan

Exclusion Criteria:

1. Subjects with a significant recent history of chronic alcohol consumption or drug addiction (past two years), or serious gastrointestinal, renal, hepatic or cardio- vascular disease, tuberculosis, epilepsy, asthma (past five years), diabetes, psychosis or glaucoma will not be eligible for this study.
2. Subjects whose clinical laboratory test values are outside the reference range may be retested at the discretion of the clinical investigator. If the clinical values are outside the range on retesting, the subject will not be eligible to participate in the study unless the clinical investigator deems the result to not be significant.
3. Subjects who have a history of allergic responses to the class of drug being tested will be excluded from the study
4. All subjects will have urine staples assayed for the presence of drugs of abuse as per of the clinical laboratory screening procedures and at each dosing period check-in. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
5. Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
6. Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate
7. Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (e.g. condom) of contraception during the course of the study (first dosing until last blood collation) or they will not be allowed to participate. Female subjects who have used hormones or contraceptives within 14 days of dosing or implanted or injected hormone contraceptives within 180 days of dosing will not be allowed to participate.
8. All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-04; Primary Completion 2004-04 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway medical research, Saint Charles, Missouri, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html